CLINICAL TRIAL: NCT06290765
Title: Efficacy and Safety of Ropeginterferon Alfa 2b (P1101) for Patients With Polycythemia Vera - A Randomized Open Label Global Multicenter Study (PARADIGM-PV)
Brief Title: Efficacy and Safety of Ropeginterferon Alfa 2b (P1101) for Patients With Polycythemia Vera
Acronym: PV
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A23-401
Record Dates: First submitted 2024-01-26; First posted 2024-03-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Polycythemia Vera; Myeloproliferative Neoplasm
Keywords: PV; MPNs; Ropeginterferon alfa-2b; P1101; Hct; Phlebotomy; JAK2
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders | interventions — Phlebotomy; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropeginterferon alfa-2b group (Experimental): Ropeginterferon alfa-2b subcutaneously (SC) every two weeks (± 3 days), target optimal dose of 500 µg.
  Interventions: Drug: Ropeginterferon alfa-2b; Procedure: Phlebotomy and aspirin
- Control group (Other): Patients will continuously receive the same therapy as s/he received for PV indication prior to screening.
  Interventions: Procedure: Phlebotomy and aspirin

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — Ropeginterferon alfa-2b subcutaneously (SC) every two weeks (± 3 days), 250 µg at Day 1, 350 µg at Week 2, and target optimal dose of 500 µg at Week 4.
  Phlebotomy should be conducted if confirmed Hct ≥48%, or confirmed Hct ≥45% that is ≥3% higher than baseline Hct value.
  Other Names: P1101
  Arms: Ropeginterferon alfa-2b group
Procedure: Phlebotomy and aspirin — Phlebotomy should be conducted if confirmed Hct ≥48%, or confirmed Hct ≥45% that is ≥3% higher than baseline Hct value, or confirmed Hct ≥45% according to the standard of care for phlebotomy at the institution regardless of the magnitude of the increase compared with the baseline. The same standard or criteria for phlebotomy eligibility should be applied for patients during the study at each study site or institution.
  Other Names: Phlebotomy and aspirin plus the other cytoreductive agents

SUMMARY:
This is a randomized, open-label, multicenter, two-arm study to assess the efficacy and safety of ropeginterferon alfa-2b for patients with PV. The entire study period is 60 weeks, including a main treatment phase (32 weeks), an extension treatment phase (24 weeks), and a safety follow-up phase (four weeks). However, the study may be extended for additional period of treatment after Week 60 pending the primary endpoint analysis at Week 32. Approximately 70 patients with PV will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of informed consent (or other age required by local regulations);
2. PV according to the World Health Organization (WHO) 2016 or 2022 Criteria;
3. At least 3 phlebotomies within 24 weeks or at least 5 phlebotomies within 52 weeks prior to screening due to inadequate control of Hct value;
4. Have the following hematological values immediately prior to randomization at baseline:

   1. Hematocrit <45%, and
   2. WBC ≥4× 109/L, and
   3. Platelets ≥100 × 109/L;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
6. Patients receiving cytoreductive therapy must be on a stable dose or minimal dose adjustments for at least 24 weeks before screening and with no planned dose change;
7. Patients who are not receiving cytoreductive therapy must have been discontinued from any prior cytoreductive therapy for at least 24 weeks before screening and have recovered from any adverse events;
8. Females of childbearing potential, as well as all women < 2 years after the onset of menopause, must agree to use an acceptable form of birth control until 60 days following the last dose of the study drug;
9. Written informed consent obtained from the patient or the patient's legal representative, and ability for the patient to comply with the study requirements.

Exclusion Criteria:

1. Patients requiring phlebotomy at Hct levels ˂45% according to Investigator judgement;
2. Clinically significant thrombosis (e.g., deep vein thrombosis or splenic vein thrombosis) or PV-related bleeding within 2 months prior to randomization;
3. Post-PV myelofibrosis as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) (Tefferi et al 2013, Barosi et al 2008);
4. Contraindication to pegylated interferon or its excipients;
5. known resistance or intolerance to interferon based therapies, as judged by Investigator;
6. Documented autoimmune disease (e.g., thyroid dysfunction, idiopathic thrombocytopenic purpura (ITP), scleroderma, psoriasis, or any arthritis of autoimmune origin). Patients with well-managed thyroid disease by oral hormonal replacement therapy could be enrolled;
7. Pulmonary infiltrates, pneumonia, and pneumonitis at screening that, in the Investigator's opinion, would jeopardize the safety or compliance with the protocol;
8. Infections with systemic manifestations, e.g., bacterial, fungal, or human immunodeficiency virus (HIV), except inactive carriers of hepatitis B (HBV) and/or hepatitis C (HCV) at screening; inactive HBV carrier is defined as the presence of HBsAg and anti-Hepatitis B e-antigen (anti-HBe) antibody, HBV DNA ˂2000 IU/ml, and normal ALT (Invernizz et al 2016); inactive HCV carrier is defined as the presence of HCV RNA but has normal ALT or with no clinically significant symptom as judged by investigator;
9. Any investigational drug less than 6 weeks prior to randomization or not recovered from the effects of prior administration of any investigational agent;
10. History or presence of depression requiring treatment with antidepressant;
11. Previous suicide attempts or at any risk of suicide at screening, in the judgement of the Investigator;
12. Any significant morbidity or abnormality which may interfere with the study participation;
13. Pregnant or lactating females;
14. History of alcohol abuse or drug abuse within the last year;
15. Evidence of severe retinopathy (e.g. cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension);
16. Significant liver (AST or ALT > 2.5 times ULN) or renal disease (creatinine > 2 mg/ml);
17. History of major organ transplantation;
18. History or presence of clinically significant neurologic diseases, e.g., uncontrolled severe seizure disorder;
19. History of malignant disease, including solid tumors and hematological malignancies (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that have been completely excised and are considered cured) within the last 3 years.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients whose Hct is maintained without phlebotomy eligibility from Week 20 through Week 32. | From Week 20 through Week 32
  Phlebotomy eligibility is defined as either: a confirmed Hct ≥45% that is at least 3% higher than the baseline Hct, a confirmed Hct ≥48%, OR a confirmed Hct ≥45% according to the standard of care for phlebotomy at the institution regardless of the magnitude of the increase compared with the baseline.